CLINICAL TRIAL: NCT05716815
Title: Prospective Randomized Study on the Efficacy of Three-dimensional Reconstructions of Bronchial and Vascular Structures on Preoperative Chest CT Scan in Patients Who Are Candidates for Pulmonary Segmentectomy Surgery
Brief Title: Prospective rAndomized sTudy efficaCy tHree-dimensional rEconstructions Segmentectomy
Acronym: PATCHES
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ospedale Centrale Bolzano (Other)
Collaborators: European Institute of Oncology (Other); Philipps University Marburg (Other); Ernst von Bergmann Hospital (Other); Chinese University of Hong Kong (Other); Wolfson Medical Center (Other Government); University of Belgrade (Other); Harvard University (Other); University of Salamanca (Other)
Responsible Party: Principal Investigator, Francesco Zaraca, MD PhD Privat Dozent, Ospedale Centrale Bolzano
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1-2023
Record Dates: First submitted 2023-01-11; First posted 2023-02-08 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Lung Cancer; Lung; Node
Keywords: Lung Segmentectomy; CT 3D Recostruction; VATS; RATS
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Intervention Model Description: A prospective multicenter randomized study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- 2D Reconstruction (Active Comparator): Before minimally invasive lung segmentectomy, preoperative chest CT scans are processed and evaluated with multi-plane (2D) reconstructions, according to the usual center protocol.
  Interventions: Diagnostic Test: CT scans 2D Reconstruction
- 2D plus 3D Reconstruction (Experimental): Before minimally invasive lung segmentectomy, preoperative chest CT scans are processed and evaluated with volume rendering (3D) reconstructions.
  Interventions: Diagnostic Test: CT scans 2D plus 3D Reconstruction

INTERVENTIONS:
Diagnostic Test: CT scans 2D Reconstruction — Before performing the surgery, patient performs a chest CT scan with contrast medium and standard two-dimensional (2D) reconstructions are performed to study the lesion, the anatomy of the bronchi and the pulmonary venous and arterial vessels.
  Arms: 2D Reconstruction
Diagnostic Test: CT scans 2D plus 3D Reconstruction — Before performing the surgery, patient performs a chest CT scan with contrast medium and standard two-dimensional (2D) reconstructions plus a 3D reconstruction are performed to study the lesion, the anatomy of the bronchi and the pulmonary venous and arterial vessels.
  Arms: 2D plus 3D Reconstruction

SUMMARY:
With this project we want to study the effectiveness of 3D reconstruction of preoperative CT to reduce operating times, blood loss and conversions after segmentectomy performed in thoracoscopy / robotics.

DETAILED DESCRIPTION:
Pulmonary segmentectomy is the surgery of first choice in malignant lung tumors with a diameter <2 cm in diameter. Patients who are candidates for this type of treatment perform usually a preoperative CT scan with two-dimensional reconstructions (2D: axial, coronary and sagittal). Today it is possible to perform a preoperative three-dimensional reconstruction (3D: volume rendering) of the vessels and bronchi using special software.

Objectives of the study is to analyze, in these patients, the benefits of 3D reconstruction of vessels and bronchi compared to 2D reconstruction, analyzing intra- and post-operative data.The study aims to randomize 288 patients over 36 months.

Study design: Prospective, randomized, controlled study. In 50% of patients the preoperative study of anatomical structures will be performed with the standard 2D method, in the remaining 50% with a 2D and 3D reconstruction. The assignment will take place through access to an online feature on the study website.

Evaluations and statistical methods The statistical analysis will be carried out using parametric and nonparametric descriptive, inferential statistical methods, while the main outcome will be carried out using the analysis of variance (ANOVA) and covariance (ANCOVA) techniques.

Ethical aspects. The study will be conducted in accordance with applicable current legislation. Approval by all relevant ethics committees will be required. Each patient will provide a written consent to participate in the study, after being properly informed.

ELIGIBILITY:
Inclusion Criteria:

* Segmentectomy performed through a minimally invasive approach (VATS or RATS).
* Pathologically proven NSCLC on the resected specimen.
* Age ≥18
* Signed written informed consent

Exclusion Criteria:

* Prior homolateral cardiothoracic surgery.
* Allergy or any other contraindication to iodinated contrast media.
* Segmentectomy performed through an open approach (thoracotomy)
* Histology different than NSCLC.
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 288 (Estimated)
Dates: Start 2023-10-01 (Estimated); Primary Completion 2026-03-01 (Estimated); Study Completion 2026-05-01 (Estimated)

PRIMARY OUTCOMES:
Conversions from minimally invasive to thoracotomic procedure | Intraoperative
  Evaluation of conversions from minimally invasive to thoracotomic procedure
Margin- and disease-free resection | 1 Month postoperative
  Margin- and disease-free resection

SECONDARY OUTCOMES:
Operating times | Intraoperative
  Evaluation of operating times
Intraoperative blood loss | Intraoperative
  Evaluation of intraoperative blood loss
Intraoperative major bleeding | Intraoperative
  Intraoperative major bleeding
Intraoperative air leaks and the use of sealants | Intraoperative
  Evaluation of intraoperative air leaks and the use of sealants
Postoperative air leaks | up to 2 weeks
  Evaluation of postoperative air leaks
Hospitalization times | up to 3 weeks
  Evaluation of hospitalization times

CONTACTS AND LOCATIONS:
Overall Officials: ZARACA FRANCESCO, Principal Investigator — Central Hospital Bolzano

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sung H, Ferlay J, Siegel RL, Laversanne M, Soerjomataram I, Jemal A, Bray F. Global Cancer Statistics 2020: GLOBOCAN Estimates of Incidence and Mortality Worldwide for 36 Cancers in 185 Countries. CA Cancer J Clin. 2021 May;71(3):209-249. doi: 10.3322/caac.21660. Epub 2021 Feb 4. PMID 33538338
- [Background] Allemani C, Matsuda T, Di Carlo V, Harewood R, Matz M, Niksic M, Bonaventure A, Valkov M, Johnson CJ, Esteve J, Ogunbiyi OJ, Azevedo E Silva G, Chen WQ, Eser S, Engholm G, Stiller CA, Monnereau A, Woods RR, Visser O, Lim GH, Aitken J, Weir HK, Coleman MP; CONCORD Working Group. Global surveillance of trends in cancer survival 2000-14 (CONCORD-3): analysis of individual records for 37 513 025 patients diagnosed with one of 18 cancers from 322 population-based registries in 71 countries. Lancet. 2018 Mar 17;391(10125):1023-1075. doi: 10.1016/S0140-6736(17)33326-3. Epub 2018 Jan 31. PMID 29395269
- [Background] Zhao ZR, Situ DR, Lau RWH, Mok TSK, Chen GG, Underwood MJ, Ng CSH. Comparison of Segmentectomy and Lobectomy in Stage IA Adenocarcinomas. J Thorac Oncol. 2017 May;12(5):890-896. doi: 10.1016/j.jtho.2017.01.012. Epub 2017 Jan 20. PMID 28111235
- [Background] Suzuki K, Saji H, Aokage K, Watanabe SI, Okada M, Mizusawa J, Nakajima R, Tsuboi M, Nakamura S, Nakamura K, Mitsudomi T, Asamura H; West Japan Oncology Group; Japan Clinical Oncology Group. Comparison of pulmonary segmentectomy and lobectomy: Safety results of a randomized trial. J Thorac Cardiovasc Surg. 2019 Sep;158(3):895-907. doi: 10.1016/j.jtcvs.2019.03.090. Epub 2019 Apr 9. PMID 31078312
- [Background] Hung MH, Cheng YJ, Chan KC, Han SC, Chen KC, Hsu HH, Chen JS. Nonintubated uniportal thoracoscopic surgery for peripheral lung nodules. Ann Thorac Surg. 2014 Dec;98(6):1998-2003. doi: 10.1016/j.athoracsur.2014.07.036. Epub 2014 Oct 28. PMID 25443006
- [Background] Wu H, Jin R, Yang S, Park BJ, Li H. Long-term and short-term outcomes of robot- versus video-assisted anatomic lung resection in lung cancer: a systematic review and meta-analysis. Eur J Cardiothorac Surg. 2021 Apr 29;59(4):732-740. doi: 10.1093/ejcts/ezaa426. PMID 33367615
- [Background] Gharagozloo F, Margolis M, Tempesta B, Strother E, Najam F. Robot-assisted lobectomy for early-stage lung cancer: report of 100 consecutive cases. Ann Thorac Surg. 2009 Aug;88(2):380-4. doi: 10.1016/j.athoracsur.2009.04.039. PMID 19632377
- [Background] Nomori H, Mori T, Shiraishi A, Fujino K, Sato Y, Ito T, Suzuki M. Long-Term Prognosis After Segmentectomy for cT1 N0 M0 Non-Small Cell Lung Cancer. Ann Thorac Surg. 2019 May;107(5):1500-1506. doi: 10.1016/j.athoracsur.2018.11.046. Epub 2018 Dec 21. PMID 30579848
- [Background] Stiles BM, Mao J, Harrison S, Lee B, Port JL, Altorki NK, Sedrakyan A. Sublobar resection for node-negative lung cancer 2-5 cm in size. Eur J Cardiothorac Surg. 2019 Nov 1;56(5):858-866. doi: 10.1093/ejcts/ezz146. PMID 31168591
- [Background] Bao F, Ye P, Yang Y, Wang L, Zhang C, Lv X, Hu J. Segmentectomy or lobectomy for early stage lung cancer: a meta-analysis. Eur J Cardiothorac Surg. 2014 Jul;46(1):1-7. doi: 10.1093/ejcts/ezt554. Epub 2013 Dec 8. PMID 24321996
- [Background] Shimizu K, Nagashima T, Ohtaki Y, Obayashi K, Nakazawa S, Kamiyoshihara M, Igai H, Takeyoshi I, Mogi A, Kuwano H. Analysis of the variation pattern in right upper pulmonary veins and establishment of simplified vein models for anatomical segmentectomy. Gen Thorac Cardiovasc Surg. 2016 Oct;64(10):604-11. doi: 10.1007/s11748-016-0686-4. Epub 2016 Jul 19. PMID 27435809
- [Background] Akiba T. Utility of three-dimensional computed tomography in general thoracic surgery. Gen Thorac Cardiovasc Surg. 2013 Dec;61(12):676-84. doi: 10.1007/s11748-013-0336-z. Epub 2013 Oct 25. PMID 24158329
- [Background] Akiba T, Marushima H, Harada J, Kobayashi S, Morikawa T. Importance of preoperative imaging with 64-row three-dimensional multidetector computed tomography for safer video-assisted thoracic surgery in lung cancer. Surg Today. 2009;39(10):844-7. doi: 10.1007/s00595-009-3965-1. Epub 2009 Sep 27. PMID 19784721
- [Background] She XW, Gu YB, Xu C, Li C, Ding C, Chen J, Zhao J. Three-dimensional (3D)- computed tomography bronchography and angiography combined with 3D-video-assisted thoracic surgery (VATS) versus conventional 2D-VATS anatomic pulmonary segmentectomy for the treatment of non-small cell lung cancer. Thorac Cancer. 2018 Feb;9(2):305-309. doi: 10.1111/1759-7714.12585. Epub 2018 Jan 3. PMID 29297974
- [Background] Xue L, Fan H, Shi W, Ge D, Zhang Y, Wang Q, Yuan Y. Preoperative 3-dimensional computed tomography lung simulation before video-assisted thoracoscopic anatomic segmentectomy for ground glass opacity in lung. J Thorac Dis. 2018 Dec;10(12):6598-6605. doi: 10.21037/jtd.2018.10.126. PMID 30746205
- [Background] Liu X, Zhao Y, Xuan Y, Lan X, Zhao J, Lan X, Han B, Jiao W. Three-dimensional printing in the preoperative planning of thoracoscopic pulmonary segmentectomy. Transl Lung Cancer Res. 2019 Dec;8(6):929-937. doi: 10.21037/tlcr.2019.11.27. PMID 32010571
- [Background] Qiu B, Ji Y, He H, Zhao J, Xue Q, Gao S. Three-dimensional reconstruction/personalized three-dimensional printed model for thoracoscopic anatomical partial-lobectomy in stage I lung cancer: a retrospective study. Transl Lung Cancer Res. 2020 Aug;9(4):1235-1246. doi: 10.21037/tlcr-20-571. PMID 32953501
- [Background] Wu Z, Huang Z, Qin Y, Jiao W. Progress in three-dimensional computed tomography reconstruction in anatomic pulmonary segmentectomy. Thorac Cancer. 2022 Jul;13(13):1881-1887. doi: 10.1111/1759-7714.14443. Epub 2022 May 18. PMID 35585765
- [Background] Oizumi H, Kanauchi N, Kato H, Endoh M, Suzuki J, Fukaya K, Sadahiro M. Anatomic thoracoscopic pulmonary segmentectomy under 3-dimensional multidetector computed tomography simulation: a report of 52 consecutive cases. J Thorac Cardiovasc Surg. 2011 Mar;141(3):678-82. doi: 10.1016/j.jtcvs.2010.08.027. Epub 2010 Sep 29. PMID 20884021
- [Derived] Zaraca F, Kirschbaum A, Pipitone MD, Bertolaccini L; PATCHES study group. Prospective randomized study on the efficacy of three-dimensional reconstructions of bronchovascular structures on preoperative chest CT scan in patients who are candidates for pulmonary segmentectomy surgery: the PATCHES (Prospective rAndomized sTudy efficaCy of tHree-dimensional rEconstructions Segmentecomy) study protocol. Trials. 2023 Sep 16;24(1):594. doi: 10.1186/s13063-023-07600-w. PMID 37717001